CLINICAL TRIAL: NCT00114309
Title: A Phase II Open-Label, Multiple-Dose Study of Intracavitary Administered 131-I-TM-601 in Adult Patients With Recurrent High-Grade Glioma
Brief Title: 131-I-TM-601 Study in Adults With Recurrent High-Grade Glioma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: TransMolecular (Industry)
Responsible Party: Susan Stewart, Vice President, Regulatory Affairs, TransMolecular, Inc.
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TM-601-002
Record Dates: First submitted 2005-06-13; First posted 2005-06-14 (Estimated); Last update posted 2009-04-03 (Estimated); Status verified 2009-04

CONDITIONS: Malignant Glioma; Glioblastoma Multiforme; GBM; Anaplastic Astrocytoma; Oligo-Astrocytoma; Gliosarcoma
Keywords: High grade recurrent glioma; Phase II; Multi-Center; Open label; Multiple dose; Brain Cancer; Brain Tumor; GBM; glioma
MeSH Terms: conditions — Glioma; Glioblastoma; Astrocytoma; Gliosarcoma; Brain Neoplasms | interventions — Chlorotoxin

ARMS (2):
- 1 (Experimental): 3 Dose Regimen
  Interventions: Drug: 131-I-TM-601
- 2 (Experimental): 6 Dose Regimen
  Interventions: Drug: 131I-TM601

INTERVENTIONS:
Drug: 131-I-TM-601 — 131I-TM601, in solution, delivered intracavitarily following surgical resection 3 weekly administrations, 0.8 mg TM601 and 40mCi 131Iodine, per dose.
  Other Names: chlorotoxin
  Arms: 1
Drug: 131I-TM601 — 131I-TM601, in solution, delivered intracavitarily following surgical resection 6 weekly administrations, 0.8 mg TM601 and 40mCi 131Iodine, per dose.
  Other Names: chlorotoxin
  Arms: 2

SUMMARY:
This drug is being developed to treat a type of brain cancer, glioma. This study was developed to evaluate the safety, time to disease progression and survival rates after treatment.

DETAILED DESCRIPTION:
This phase II trial was designed in two sequences. The first sequence, which is now complete to accrual was an open-label, dose escalation, multi-dose study and treated 12 evaluable patients with high-grade glioma.

The second sequence is currently open and accruing eligible subjects with high-grade glioma. The trial is an open-label, randomized study and will accrue a total of 54 evaluable patients. Eligible subjects will be randomized to receive either 3 or 6 injections of 131-I labeled TM-601 (131-I-TM-601), in weekly intervals at the dose determined in the first sequence of the trial. Patients will undergo debulking surgery and placement of a ventricular access device into the tumor cavity for administration of 131I-TM-601. Patients who participated in the first sequence are not eligible to participate in the second sequence of the study.

High-grade gliomas include; glioblastoma multiforme, anaplastic astrocytoma, oligoastrocytoma or gliosarcoma.

Patients will undergo follow-up clinical examinations and magnetic resonance imaging (MRI) assessments, at defined intervals, until 12 months after the first study dose.

ELIGIBILITY:
Inclusion Criteria:

* Patient must have a histologically confirmed unilateral, supratentorial malignant glioma (grade 3 or 4, anaplastic astrocytoma, gliosarcoma, glioblastoma multiforme or malignant oligoastrocytoma)
* Patient must have glioma progression or recurrence following radiotherapy that was no less than 50 Gy (+/- chemotherapy; +/- surgery)
* Patient must be a candidate for resection of the recurrent tumor (surgical requirements are detailed in the study protocol)
* Imaging must show recurrent, unilateral, supratentorial tumor(s)
* There is no diffuse leptomeningeal disease
* For patients with previous radiosurgery or enhanced radiotherapy, based on neurosurgeon's judgment, the area of enhancement can be removed during the surgery
* Patient must have recovered from toxicity of prior therapy
* Patient must be > 18 years of age.
* Patient has a Karnofsky Performance Status greater than or equal to 60%
* Patient must have a life expectancy of at least 3 months
* Patient has no uncontrolled seizures or other neurological conditions which would interfere with evaluation
* Patient is not currently receiving, or is not anticipated to receive, concomitant anticancer agent(s) during the course of this study
* Patient must have given informed consent

Exclusion Criteria:

* Patient with concurrent malignancy (except curatively treated basal or squamous cell carcinoma of the skin or carcinoma in situ of cervix and/or breast) or patients with prior malignancies that have not been disease-free for five years
* Patient has presence of non-contiguous satellite lesions
* Patient with known allergy to iodine, iodine containing drugs or contrast agent
* Patient with the potential for pregnancy or impregnating their partner and who do not agree to follow an acceptable birth control method to avoid conception
* Pregnant or breast feeding females
* Patient is not maintained on a stable corticosteroid regimen
* New onset of conditions not present prior to surgery (as detailed in Study Protocol) which would make patient an inappropriate study candidate, or as determined by Investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2004-11; Primary Completion 2009-03 (Actual); Study Completion 2009-08 (Estimated)

PRIMARY OUTCOMES:
Determine Maximum Tolerated Dose (MTD) of 131-I-TM-601 administered intracavitary to patients with recurrent high-grade glioma | 28 days post last dose
Determine the toxicity of a three (3) and six (6) dose cycle of 131-I-TM-601 administrations into the tumor resection site of patients with recurrent high-grade glioma | 28 days post last dose and then at 3 month intervals from first dose, until disease progression
Evaluate the 6 and 12-month rate of progression and survival of patients with recurrent high-grade glioma treated with a three (3) or six (6) dose cycle of 131-I-TM-601 | at 3 month intervals from first dose administration, until disease progression
Evaluate the overall time to progression and death of patients with recurrent high-grade glioma treated with either a three (3) or six (6) dose cycle of 131-I-TM-601 | at 3 month intervals until disease progression

SECONDARY OUTCOMES:
Evaluate if either a three (3) or six (6) dose cycle of 131-I-TM-601 affects Quality of Life | 3 month intervals until disease progression

CONTACTS AND LOCATIONS:
Overall Officials: John Fiveash, MD, Principal Investigator — University of Alabama at Birmingham
Locations (19):
- United States (19):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - City of Hope, Duarte, California
  - Cedars-Sinai Medical Center, Los Angeles, California
  - Florida Hospital Cancer Institute, Orlando, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - Emory University, Atlanta, Georgia
  - Northwestern University, Chicago, Illinois
  - University of Chicago, Chicago, Illinois
  - Johns Hopkins Medical Center, Baltimore, Maryland
  - Tufts-New England Medical Center, Boston, Massachusetts
  - Henry Ford Hospital, Detroit, Michigan
  - Lacks Cancer Center at St. Mary's Health Care, Grand Rapids, Michigan
  - St. Louis Hospital, St Louis, Missouri
  - Washington University Medical Center, St Louis, Missouri
  - Columbia University Medical Center, New York, New York
  - Carolina Neurosurgery and Spine, Charlotte, North Carolina
  - Mary Crowley Medical Research Center, Dallas, Texas
  - Huntsman Cancer Institute, Salt Lake City, Utah
  - University of Washington, Seattle, Washington

REFERENCES:
- [Background] Mamelak AN, Jacoby DB. Targeted delivery of antitumoral therapy to glioma and other malignancies with synthetic chlorotoxin (TM-601). Expert Opin Drug Deliv. 2007 Mar;4(2):175-86. doi: 10.1517/17425247.4.2.175. PMID 17335414
- [Background] Lyons SA, O'Neal J, Sontheimer H. Chlorotoxin, a scorpion-derived peptide, specifically binds to gliomas and tumors of neuroectodermal origin. Glia. 2002 Aug;39(2):162-73. doi: 10.1002/glia.10083. PMID 12112367
- [Result] Mamelak AN, Rosenfeld S, Bucholz R, Raubitschek A, Nabors LB, Fiveash JB, Shen S, Khazaeli MB, Colcher D, Liu A, Osman M, Guthrie B, Schade-Bijur S, Hablitz DM, Alvarez VL, Gonda MA. Phase I single-dose study of intracavitary-administered iodine-131-TM-601 in adults with recurrent high-grade glioma. J Clin Oncol. 2006 Aug 1;24(22):3644-50. doi: 10.1200/JCO.2005.05.4569. PMID 16877732
- [Result] Hockaday DC, Shen S, Fiveash J, Raubitschek A, Colcher D, Liu A, Alvarez V, Mamelak AN. Imaging glioma extent with 131I-TM-601. J Nucl Med. 2005 Apr;46(4):580-6. PMID 15809479